CLINICAL TRIAL: NCT04688424
Title: Functional Electrical Stimulation Assisted Cycling to Improve Fitness and Strength in Children With Cerebral Palsy
Brief Title: FES Assisted Cycling in Children With CP
Acronym: CP FES Cycling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Collaborators: Shriners Hospitals for Children (Other)
Responsible Party: Principal Investigator, Samuel C.K. Lee, PhD, PT, Principal Investigator, Associate Professor, Dept of Physical Therapy, University of Delaware
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5R01HD062588-02 (NIH)
Record Dates: First submitted 2015-05-15; First posted 2020-12-30 (Actual); Last update posted 2020-12-30 (Actual); Status verified 2020-12

CONDITIONS: Cerebral Palsy Spastic Diplegia
Keywords: Cerebral Palsy; Functional electrical stimulation; Cycling
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- FES + Cycling (Experimental): Functional electrical stimulation cycling group
  Interventions: Device: FES; Other: Cycling
- Cycling only (Active Comparator): Volitional cycling group (no electrical stimulation)
  Interventions: Other: Cycling
- Control (No Intervention): control group

INTERVENTIONS:
Device: FES — FES will be applied via surface electrodes placed over bilateral quadriceps muscles. FES-stimulation will be ramped from sensory level (the level at which the individual feels a cutaneous sensation from the stimulation) to the maximum-tolerated level using a closed loop system controlled by computer software Subjects will exercise at home, three times per week, with FES on for 8 weeks with a goal of attaining 30 minutes of continuous cycling per session. If the individuals are unable to cycle for 30 continuous minutes, rest breaks will be provided with a goal of cycling for a total of 30 minutes. The length of each session will be approximately 45 minutes, with 15 minutes of set-up and 30 minutes of cycling.
  Arms: FES + Cycling
Other: Cycling — Subjects will exercise at home, three times per week, without FES for 8 weeks with a goal of attaining 30 minutes of continuous cycling per session. If the individuals are unable to cycle for 30 continuous minutes, rest breaks will be provided with a goal of cycling for a total of 30 minutes. The length of each session will be approximately 45 minutes, with 15 minutes of set-up and 30 minutes of cycling.
  Arms: Cycling only; FES + Cycling

SUMMARY:
This project proposes to assess if Functional Electrical Stimulation (FES) assisted cycling can improve the cycling ability, muscle strength, cardiovascular health, quality of life, self perception and functional mobility of adolescents with CP better than a volitional cycling program or a non-intervention control group.

DETAILED DESCRIPTION:
Aim 1: To compare the effects of 8-weeks of FES-assisted cycling training on improving cardiorespiratory fitness, walking function, self-motivated exercise/recreation, self-perception and functional mobility and quality of life of adolescents with spastic CP with marginal walking ability (Gross Motor Function Classification System Levels II - IV) vs. 8-weeks of volitional cycling training and a non-intervention control group.

Aim 2: To compare the effects of 8-weeks FES-assisted cycling training on changes in cycling ability of adolescents with spastic CP with marginal walking ability vs. 8-weeks of volitional cycling training and a nonintervention control group.

Aim 3: To elucidate the mechanisms for potential improvements in cycling ability after 8-weeks of FES-assisted or volitional cycling training of adolescents with spastic CP and marginal walking ability.

ELIGIBILITY:
Inclusion Criteria:

* Spastic CP (di-, tetra-, or triplegic)
* Level II, III or IV GMFCS classification
* Sufficient covering of the femoral head in the acetabulum (migration % < 40)
* Adequate range of motion of the hips, knees and ankles to allow pedaling
* Visual, perceptual, cognitive, and communication skills to follow multiple step commands for attending to exercise and data collection
* Seizure-free or well controlled seizures

Exclusion Criteria:

* Athetoid, ataxic, or hemiplegic CP
* Significant scoliosis (primary curve > 40°)
* Spinal fusions extending into the pelvis
* Severe tactile hypersensitivity
* Joint instability or dislocation in LE
* LE surgery or fractures in the past year
* Botox injections to LE in the past 6 months
* Severe spasticity in LE (Mod Ashworth 4)
* LE joint pain during cycling
* Hx of pulmonary disease limiting exercise tolerance or Hx of cardiac disease
* Severely limited ROM / contractures that prevent the subject from being able to be safely positioned on the cycle
* Pregnancy

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 39 (Actual)
Dates: Start 2008-04; Primary Completion 2016-06-30 (Actual); Study Completion 2016-06-30 (Actual)

PRIMARY OUTCOMES:
Change in cycling Ability | Outcome assessed: Pre Training (week 0), Mid Training (week 4), Post Training (week 8), Follow-Up (week 16)
  Change in cycling cadence from pre-training to post-training and at follow-up will be assessed.
Change in Energy Expenditure | Outcome assessed: Pre Training (week 0), Mid Training (week 4), Post Training (week 8), Follow-Up (week 16)
  Energy expenditure is a measure of cardiovascular fitness. Change in energy expenditure from pre-training to post-training and at follow-up will be assessed.
Change in Gait speed | Outcome assessed: Before Training (week 0), Mid Training (week 4), After Training (week 8), Follow-Up (week 16)
  Gait speed will be measured using a GAITRite Portable Walkway System (CIR Systems Inc; Havertown, PA). We will measure the change in gait speed from pre-training to post-training and at follow-up.
Change in Spatiotemporal gait parameter | Outcome assessed: Before Training (week 0), Mid Training (week 4), After Training (week 8), Follow-Up (week 16)
  Step length will be measured using a GAITRite Portable Walkway System (CIR Systems Inc; Havertown, PA). We will measure the change in step length from pre-training to post-training and at follow-up.
Change in Muscle Strength | Outcome assessed: Before Training (week 0), Mid Training (week 4), After Training (week 8), Follow-Up (week 16)
  Isometric maximum voluntary exertion testing of hip extensors & flexors, knee extensors & flexors, and ankle plantarflexors. We will measure the change in isometric maximum voluntary exertion from pre-training to post-training and at follow-up.
Change in Walking Distance | Outcome assessed: Before Training (week 0), Mid Training (week 4), After Training (week 8), Follow-Up (week 16)
  6 minute walk test (6MWT) measures walking distance. Walking distance (in a fixed period of time) is an indicator of endurance. We will measure the change in walking distance from pre-training to post-training and at follow-up.
Change in Timed Up-And-Go | Outcome assessed: Before Training (week 0), Mid Training (week 4), After Training (week 8), Follow-Up (week 16)
  Timed Up-And-Go (TUG) is a measure of functional mobility and will allow for assessing the impact of anticipated improvements in motor control and gait biomechanics. We will measure the change in TUG test from pre-training to post-training and at follow-up.
Change in Pedometer measurement | Outcome assessed: Before Training (week 0), Mid Training (week 4), After Training (week 8), Follow-Up (week 16)
  Pedometer measurements to allow an unbiased report of the subject's activity level at home and in the community. We will measure the change in pedometer measurements from pre-training to post-training and at follow-up.
Change in Electromyography | Outcome assessed: Before Training (week 0), Mid Training (week 4), After Training (week 8), Follow-Up (week 16)
  Muscle activation timing measured with electromyography (EMG) during analysis allows for mechanistic study of anticipated improvements in motor control as well as comparison to typical norms. We will measure the change in EMG from pre-training to post-training and at follow-up.
Change in Self-Assessment | Outcome assessed: Before Training (week 0), Mid Training (week 4), After Training (week 8), Follow-Up (week 16)
  Canadian Occupational Performance Measure (COPM) is a 10 point scale to rate one's own level of performance and satisfaction with performance. 1 mean poor performance low satisfaction and 10 means very good performance high satisfaction. We will measure the change in COPM scores from pre-training to post-training and at follow-up.
Change in Health related Quality of Life | Outcome assessed: Before Training (week 0), Mid Training (week 4), After Training (week 8), Follow-Up (week 16)
  The KINDL questionnaire is administered to measure changes in health-related quality of life. The questionnaire is completed by the adolescent and a caregiver. The KINDL standard scale and "Disease Module" is administered. The standard scale contains 24 items comprised of Physical, Emotional, Self-Esteem, Family, Friends and School sub-scales. The 6-item "Disease Module" that measures the child's and caregiver's perceptions about CP. Scores for each item ranges from 1-5. The total score is the sum of all item scores, transformed to a 0-100 scale. Higher scores indicate better quality of life. We will measure the change in KINDL scores from pre-training to post-training and at follow-up.
Change in Self-Perception | Outcome assessed: Before Training (week 0), Mid Training (week 4), After Training (week 8), Follow-Up (week 16)
  Self-Perception (Piers-Harris-2) survey measures physical and emotional well-being and self-esteem and will allow assessment of the impact of anticipated improvements in motor control and gait biomechanics from training. We will measure the change in Piers-Harris scores from pre-training to post-training and at follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Lee, PT, PhD, Principal Investigator — Physical Therapy Department, University of Delaware
Locations (1):
- Shriners Hospitals fof Children, Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
The proposed experiments will generate data for publications in high quality peer reviewed journals. We will also present our findings at national meetings of neurorehabilitation scientists and clinicians and neuroscience and motor control meetings. To have the most impact, it is important that we present our findings to both clinicians and scientists, therefore, in addition to these standard approaches, we will seek out regular opportunities to present both the rationale and results of our work to local and regional clinicians as well as local and regional stroke support groups.
Supporting Information: Study Protocol
Time Frame: Following publication of primary results.

REFERENCES:
- See also: Dr. Lee's research studies — https://sites.udel.edu/pt/research/samuel-lee-pt-mpt-phd/